CLINICAL TRIAL: NCT05592678
Title: Novel Methods for Clinical Trials in Dementia and Cognitive Decline
Brief Title: δ in Dementia Clinical Trials
Acronym: δND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Donald Royall, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20220551H; R01AG080548 (NIH)
Record Dates: First submitted 2022-10-13; First posted 2022-10-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease (AD); Dementia; Cognitive Decline; Mild Cognitivie Impairment (MCI)
Keywords: adipokines; cognition; dementia; functional status; intelligence
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction | interventions — Donepezil

STUDY DESIGN:
Intervention Model Description: a double-blind group assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blind to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Predicted Responders (Other): Group assignment determined by a response predictor algorithm derived from remotely acquired caregiver reports of cognitive performance. The donepezil administered during the study is prescribed by the subject provider as standard of care.
  Interventions: Other: Donepezil
- Predicted Non-Responders (Other): Group assignment determined by a response predictor algorithm derived from remotely acquired caregiver reports of cognitive performance. The donepezil administered during the study is prescribed by the subject provider as standard of care.
  Interventions: Other: Donepezil

INTERVENTIONS:
Other: Donepezil — Donepezil is administered as a standard of care treatment by the subject's provider.
  Other Names: Aricept ®

SUMMARY:
The goal of this clinical trial is to demonstrate potential improvements in clinical trial methods relating to dementia and cognitive decline. The main questions it aims to answer are:

* Can an intervention's outcome be better assessed by a latent variable ("δ") integrating cognitive performance with functional status?
* Can latent biomarkers of δ guide the selection of an intervention that will modulate dementia severity?
* Can a latent variable, derived from information collected remotely from caregivers, preselect subjects most likely to respond to the intervention?
* Is the effect of the intervention in fact medicated by changes in the targeted biomarker?

In this case, the biomarker will be a latent variable derived from several proteins measured in blood (i.e., so-called "adipokines"). The intervention will be donepezil, a medication approved for the treatment of Alzheimer's Disease, but only recently associated with adipokine changes.

Participants with cognitive impairment and their caregivers will be interviewed by telephone and those newly prescribed donepezil by their provider for cognitive impairment will be recruited and enrolled. On the basis of the caregiver's report, the cognitively impaired subjects will be assigned to two groups based on a prediction of their response to donepezil. Researchers will compare those groups to see if dementia severity, as measured by δ, improves in predicted responders, and whether the change in the d-score is mediated by changes in adipokines.

DETAILED DESCRIPTION:
Title: "Novel Methods for Clinical rials in Dementia and Cognitive Decline"

Study Description: This is a double-blind assignment clinical study to test novel approaches to clinical trial methods. 1) The study team will pre-select cases most likely to benefit from adipokine modulation by a telephone assessment. 2) The study team will pre-select subjects with clinical and preclinical dementia most likely to respond to therapy. 3) The study team will test the drug donepezil's effect on dementia severity, in predicted responders and non-responders, as measured by a latent dementia phenotype "δ' and 4) test a latent Adipokines biomarker construct as a mediator of their association in the predicted responders.

Objectives:

Primary Objective: To assess donepezil's effect on dementia severity as measured by δ in LOI subgroups and across LOI subgroups.

Secondary Objective: To test Adipokines as a mediator of donepezil's effect on dTEL.

Tertiary/Exploratory: To test whether donepezil reverses dementia in cases preselected to by "LOI" analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory outpatient volunteers with competent informants. Competent informants are cognitively normal individual(s) who interacts with the person on a regular (at least 5 or more hours/week) basis and in the opinion of the PI can provide adequate collateral information on the participant's memory and cognitive status.
2. Aged 65-100 years
3. Clinical diagnosis of AD, or MCI.
4. Capacity to give informed consent. If a patient is found to clinically decline during the course of the study and no longer able to provide consent, continued participation will be evaluated by the PI on a case-by-case basis.
5. GDS score (15 item) ≤ 6.
6. No significant visual or hearing impairments
7. A standardized dECog score between 1.5 and 3.5 relative to ADNI's cohort.
8. Assignment to "Group 1" by a LOI assessment of Adipokine adjusted v. unadjusted dECog scores.
9. In the opinion of the participant's physician, Donepezil is medically indicated for the treatment of memory impairment and the participant has obtained a prescription for it. .
10. Physician instructions are in line with a titration to a dosage of 10 mg Qd per the standard dosing guidelines for Donepezil. If participant not able to tolerate 5 mg titration over 4 weeks, PI will need to authorize continued enrollment.

Exclusion Criteria:

1. A history of psychosis, including visual hallucinations;
2. History or treatment for Parkinson's, or tremor, or Rapid Eye Movement (REM) behavior disorder;
3. History or treatment for atrial fibrillation;
4. History of bradycardia or syncopal events;
5. Chronic diarrhea, h/o colonic resection or irritable bowel syndrome;
6. Treatment for cancer in the last 5 years (excluding skin cancers);
7. Major surgery in the last year;
8. Treatment for a seizure disorder with anticonvulsants
9. Current treatment with donepezil or any other AChEI or exposure within the last year.
10. Treatment with opiates, muscle relaxants, or systemic steroids.
11. In the opinion of the PI, treatment with AChEI is not appropriate due to a possible negative risk/benefit ratio based on past medical history or endorsement of symptoms during the screening interview.
12. In the opinion of the treating physician, the patient must begin therapy with AChEI immediately due to any delays having an unacceptable impact on the patient's QoL.
13. Co-participation in another study that the PI feels would pose a safety risk or adversely affect data integrity of this study.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
dTEL change | At baseline, and weeks 4, 12 and 24.
  Change in a latent dementia-specific phenotype derived from cognitive assessment.

SECONDARY OUTCOMES:
ADIPOKINES change | Baseline and week 24.
  Change in a latent construct derived from eight "Adipokine" proteins measured in blood.

OTHER OUTCOMES:
Dementia "Reversion" | Week 24
  The frequency of dementia "reversion" defined as a final dTEL score > -0.40, i.e., the optimal d-score that discriminates subjects with AD from those with MCI in the Alzheimer's Disease Neuroimaging Initiative (ADNI).

CONTACTS AND LOCATIONS:
Overall Officials: Donald R. Royall, MD, Principal Investigator — University of Texas
Locations (1):
- Univeristy of Texas Health Science Center at San Antonio (UTHSCSA), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers 5 years after the completion of the primary endpoint by contacting royall@uthscsa.edu
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers 5 years after the completion of the primary endpoint by contacting royall@uthscsa.edu